CLINICAL TRIAL: NCT05556876
Title: Effect of Oral Nutritional Supplements on Muscle Strength in Older Patients at Nutritional Risk Discharged With a Rehabilitation Plan
Brief Title: Effect of Oral Nutritional Supplements to Older Patients Discharged With a Rehabilitation Plan
Acronym: NUTRIMUSCLE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Nutricia, Inc. (Industry)
Responsible Party: Principal Investigator, Anne Marie Beck, Senior researcher, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: version2/30.03.2022
Record Dates: First submitted 2022-09-21; First posted 2022-09-27 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Nutritional Risk; Rehabilitation; Oral Nutritional Supplements
Keywords: muscle strenght; quality of life; body composition; protein intake

STUDY DESIGN:
Intervention Model Description: A single-blinded randomised study
Who Masked: Outcomes Assessor
Masking Description: two set of files
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): the intervention group will be provided with oral nutritional supplements for 12 weeks after discharge
  Interventions: Dietary Supplement: Protein omega-3
- Control (No Intervention): the control group will receive usual care after discharge

INTERVENTIONS:
Dietary Supplement: Protein omega-3 — An oral supplement with a high content of protein and with essential fatty acids
  Arms: Intervention

SUMMARY:
The purpose of the study is to investigate whether an extra intake of energy and protein in the form of nutritional drinks twice a day for 12 weeks can improve muscle strength, muscle mass, quality of life and the implementation of rehabilitation in elderly patients at nutritional risk who are discharged to municipal rehabilitation

DETAILED DESCRIPTION:
The study is a single-blind randomised study where the subjects will be randomly divided into two groups. A group that must consume nutritional drinks in connection with their rehabilitation and a group that must do nothing extra. Based on a statistical power calculation, we will include a total of 124 patients.

In connection with the experiment, different data will be collected three times, in connection with the discharge from the hospital, after 6 weeks via the telephone and after 12 weeks. During a home visit. Here, various questionnaires will have to be answered and data on muscle strength and muscle mass will be collected. Further CRP, vitamin D status and EPA/DHA content in blood will be assessed.

In addition, data is collected from the patient's medical record about e.g. readmissions

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 65 years old
* Independent stand function

  * Able to speak and understand Danish
  * At nutritional risk according to NRS-2002
  * (Expected to be) discharged with a new rehabilitation plan
  * Admitted to the medical and orthopaedic departments of Gentofte or Herlev Hospital

Exclusion Criteria:

* Active cancer

  * Renal insufficiency (eGFR < 27 mL/min/1.73m2)
  * Cognitive impairment (not able to comprehend the purpose of the study/give informed consent)
  * Terminal disease
  * Exclusively receiving texture modified food, enteral or parenteral nutrition
  * Planning to lose weight/go on a special diet
  * Planned transfer to other hospitals/departments
  * Pacemaker/other implanted electrical stimulants (due to Bio-Impedance Analysis (BIA)

    * Taking fish-oil supplements as a medical prescription due to hypertriglyceridemia
    * Taking fish-oil supplements for other reasons and do not wish to stop this during the study period

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Leg Muscle strength | change from baseline to 12 weeks follow-up
  Chair stand

SECONDARY OUTCOMES:
Hand grip Muscle strength | change from baseline to 12 weeks follow-up
  Hand grip strength
Health related quality of life | Change from baseline to 6 and 12 weeks follow-up
  EQ5D5L questionnaire with five dimensions and five level of answers. To be converted to an index were -1 is worst and 1 is best health related quality of life
Activities of daily living | Change from baseline to 6 and 12 weeks follow-up
  Functional recovery score The eleven-item questionnaire is comprised of three main components: basic activities of daily living (BADL) assessed by four items, instrumental activities of daily living (IADL) assessed by six items, and mobility assessed by one item. Basic activities of daily living comprise 44 percent of the score; instrumental activities of daily living comprise 23 percent, and mobility comprises 33 percent. Complete independence in basic and instrumental activities of daily living and mobility results in a score of 100 percent
energy and protein intake | at 12 weeks follow-up
  24 hour dietary recall
Appetite | Change from baseline to 12 week follow-up
  Simplified Nutritional Appetite Questionnaire [SNAQ. The questionnaire results in a score ranging from 5 to 20, where 5 is lowest appetite
Muscle mass | Change from baseline to 12 week follow-up
  Calf circumference assessment of muscle mass
Frailty | Change from baseline to 12 weeks follow-up
  The "FRAIL" Questionnaire includes questions concerning Fatigue, Resistance (capability of stair climbing),Aerobic( walking distance), Illnesses (multi morbidity), and Loss of weight. Physical frailty, pre-frailty and non-frailty is defined as having 3 or greater; 1 or 2 or no factors respectively
initiation and completion of rehabilitation | at 12 week follow-up
  questionnaire were participants can document their attendance to exercise rehabilitation and reasons for not attending.
compliance to oral nutritional supplements | at 12 weeks follow-up
  a diary were participants can register their intake of supplements and eventual side effects. A compliance of 100% is aimed for as optimal
readmissions | 30 days and 38 weeks after discharge
  number, length and percentage of readmissions after discharge will be calculated
mortality | 30 days and 38 weeks after discharge
  number and percentage of mortality after discharge will be calculated
inflammation | change from baseline to 12 weeks follow-up
  blood measurements of CRP and omega-3 fatty acids
vitamin D status | change from baseline to 12 weeks follow-up
  blood measurements of vitamin D
Hydration status | Change from Baseline to 12 weeks follow up
  Blood measurements and calculation of serum osmolarity

CONTACTS AND LOCATIONS:
Overall Officials: Tina Munk, PhD, Study Director — Herlev and Gentofte Hospital
Locations (1):
- Herlev and Gentofte hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jensen A, Ninh ED, Tetens I, Beck AM. Oral nutritional supplements for older hip fracture patients at nutritional risk (NUTRI-MUSCLES)-a feasibility trial for a two-armed RCT. Pilot Feasibility Stud. 2026 Jan 21. doi: 10.1186/s40814-026-01763-4. Online ahead of print. PMID 41566545